CLINICAL TRIAL: NCT00897962
Title: Serum Glycan Analysis in Breast Cancer
Brief Title: Blood Glycan Biomarkers in Women With Stage IV Breast Cancer
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 234870; UCD-186; UCD-200614601; CDR0000583066 (Other: UC Davis)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Metastatic Breast Cancer: Patients with metastatic breast cancer receiving treatment with chemotherapy, endocrine therapy or targeted therapy
  Interventions: Other: Metastatic Breast Cancer
- Non-cancer medical illness: Patients with non-cancer medical condition
  Interventions: Other: Non-cancer medical illness
- Healthy Controls: Healthy patients being seen for an annual exam
  Interventions: Other: Healthy Controls

INTERVENTIONS:
Other: Healthy Controls — One blood draw (2 teaspoons)
  Groups: Healthy Controls
Other: Metastatic Breast Cancer — Blood samples will be drawn every 3 months, for up to 18 months.
  Groups: Metastatic Breast Cancer
Other: Non-cancer medical illness — One blood draw (2 teaspoons)
  Groups: Non-cancer medical illness

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur and identify biomarkers related to cancer.

PURPOSE: This research study is looking at blood glycan biomarkers in women with stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To profile serum glycan biomarkers in women with metastatic stage IV breast cancer, healthy controls, and patients with noncancer medical illness.
* To determine whether serial serum glycan biomarkers correlate with response of metastatic disease to treatment.

OUTLINE: This is a multicenter study.

Blood is collected from patients with metastatic breast cancer, patients with noncancerous illness, and healthy volunteers. Samples are analyzed for serum glycan biomarkers by matrix-assisted laser desorption/ionization (MALDI) and Fourier transform ion-cyclotron resonance mass spectrometry (FT ICR MS) methods.

Blood samples are collected every 3 months for up to 18 months from patients with metastatic breast cancer. Patients without cancer have a single sample collected.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patient or participant at the Women's Health Clinic, the Internal Medicine Clinic, or at the UC Davis Cancer Center, meeting 1 of the following criteria:

  * Diagnosis of stage IV metastatic breast cancer, receiving active treatment with chemotherapy, endocrine therapy, or targeted therapy
  * Patients/participants without cancer

    * Healthy control being seen for annual exams, meeting the following criteria:

      * No chronic disease
      * Not on regular prescribed medications
    * Patient without cancer being seen in the Internal Medicine Clinic
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Not pregnant or breast feeding
* No other active cancer

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic breast cancer receiving active chemotherapy, endocrine therapy or targeted therapy Healthy age matched controls without chronic diseases and not on regular prescription medications Patients seen at Internal Medicine Clinic for any reason other than active, metastatic cancer
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2006-09; Primary Completion 2011-02 (Actual); Study Completion 2016-01-12 (Actual)

PRIMARY OUTCOMES:
Profiling serum glycan biomarkers in patients with metastatic breast cancer, healthy controls, and patients with noncancer medical illness | up to 18 months

SECONDARY OUTCOMES:
Predictability of serial serum biomarkers in determining disease response and/or progression | Up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Helen K. Chew, MD, Study Chair — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States